CLINICAL TRIAL: NCT01336270
Title: Characterisation of T Lymphocytes, NK Cells and Macrophages in Melanoma Patients: Impact on Immunity Versus Immunosuppression
Brief Title: Characterisation of T Lymphocytes, NK Cells and Macrophages in Melanoma Patients
Acronym: IMMUMELA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P090405
Record Dates: First submitted 2011-04-14; First posted 2011-04-15 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: Melanoma; NK cells; T lymphocytes; macrophages
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A bank of biological samples (human plasma and cells) will be done
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- MELANOMA 10mm: patients with a melanoma larger than 10mm or with cutaneous metastasis
  Interventions: Other: biological collection
- STAGE III MELANOMA: stage III melanoma patients who shall undergo a regional lymph node dissection
  Interventions: Other: biological collection
- SENTINEL NODE PROCEDURE: retrospective study of patients who underwent a sentinel node procedure
  Interventions: Other: biological collection
- STAGE IV MELANOMA: stage IV patients achieves of inoperable melanomas the stage(stadium) III or IV that must receive in treatment(processing) a chemotherapy (by the dacarbazine or by the cisplatin or by the inhibitor of B-raf) and carrier of at least two cutaneous metastases
  Interventions: Other: biological collection

INTERVENTIONS:
Other: biological collection — to collect some human cell samples in melanoma
  Other Names: to collect some human cell samples in melanoma

SUMMARY:
Melanoma tumor tissue ( in particular regressive areas) present a lymphocytic infiltrate with an anti-tumoral specificity. The aim of the study is to analyse at different stages of the disease, tumor samples and to characterise the cellular infiltrate in situ ( in particular T lymphocytes, NK cells and macrophages), the role of inhibitor receptors on in situ immunosuppression, and potential modulation by medical treatments such as dacarbazine.

DETAILED DESCRIPTION:
The study is divided in 4 parts:

Part 1: study of cellular infiltrate (lymphocytes) performed on large primary melanoma and cutaneous metastasis ( fresh samples) Part 2: NK cells study on metastatic regional lymph nodes ( fresh samples) and blood samples Part 3: a retrospective study of macrophages in sentinel lymph nodes and in corresponding primary melanomas Part 4: study of the cellular modulation by the chemotherapy (DTIC or cisplatin or inhibitor of B-raf) which(who) will be made on two cutaneous metastases by patient (one taken before the treatment(processing) and one taken during the evaluation after 2 or 3 cycles of treatment(processing))

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed melanoma-patients informed of the aims of the study , the modalities
* Patients who signed the consent form ou a non opposition form signed by the patient or by a relative

According to study part:

Part 1: patients with a melanoma larger than 10mm or with cutaneous metastasis Part 2: stage IV melanoma patients who shall undergo a regional lymph node dissection Part 3: retrospective study of patients who underwent a sentinel node procedure Part 4: Patients achieves of inoperable melanomas the stage(stadium) III or IV that must receive in treatment (processing) a chemotherapy (by the dacarbazine or by the cisplatin or by the inhibitor of B-raf) and carrier of at least two cutaneous metastases

Exclusion Criteria:

* Refusal to take part in the study (patient or relative)
* Contraindications known to the xylocaine (groups 1,2, and 4)
* No affiliated to the social security system (groups 1, 2, and 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1: patients with a melanoma larger than 10mm or with cutaneous metastasis Part 2: stage III melanoma patients who shall undergo a regional lymph node dissection Part 3: retrospective study of patients who underwent a sentinel node procedure Part 4: stage IV Patient achieves of inoperable melanomas the stage(stadium) III or IV that must receive in treatment(processing) a chemotherapy (by the dacarbazine or by the cisplatin or by the inhibitor of B-raf) and carrier of at least two cutaneous metastases
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Impact of cellular infiltrate - Group 1 | 2 years
  Impact of cellular infiltrate on disease free survival at 2 years
Impact of NK cell infiltrate - Group 2 and 3 | 2 and 3 years
  Impact of NK cell infiltrate in metastatic lymph node on disease free survival and overall survival at 2 and 3 years
Modifications of cellular infiltrate - Group 4 | 2 months
  Modifications of cellular infiltrate after chemotherapy (after 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Françoise Avril, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Messaoudene M, Perier A, Fregni G, Neves E, Zitvogel L, Cremer I, Chanal J, Sastre-Garau X, Deschamps L, Marinho E, Larousserie F, Maubec E, Avril MF, Caignard A. Characterization of the Microenvironment in Positive and Negative Sentinel Lymph Nodes from Melanoma Patients. PLoS One. 2015 Jul 28;10(7):e0133363. doi: 10.1371/journal.pone.0133363. eCollection 2015. PMID 26218530